CLINICAL TRIAL: NCT07343947
Title: Melatonin Supplementation in Ovarian Response: a Double-blind Randomized Controlled Trial on Follicular Fluid Melatonin Levels and Reproductive Outcomes in Infertile Women
Brief Title: Melatonin Supplementation in Ovarian Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Jose Maria Soares Junior, Head of Gynecology Department, Principal Investigator, Clinical Professor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CEP-USP No. 4,996,660
Record Dates: First submitted 2025-12-02; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Infertility; Infertility (IVF Patients); Infertile Women Undergoing IVF or ICSI
Keywords: IVF; Infertile women; Melatonin; follicular fluid; ovarian response
MeSH Terms: conditions — Infertility | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator)
  Interventions: Other: Sham (No Treatment)
- Melatonin suplementation (Experimental)
  Interventions: Drug: 5mg melatonin supplementation

INTERVENTIONS:
Drug: 5mg melatonin supplementation — 5 mg melatonin suplementation
  Arms: Melatonin suplementation
Other: Sham (No Treatment) — Sham (no treatment)
  Arms: Control

SUMMARY:
Melatonin is a potent antioxidant, has been proposed to improve ovarian response and oocyte quality in assisted reproductive technologies (ART). This study evaluated the effects of melatonin supplementation on follicular fluid melatonin levels, hormonal profiles, and reproductive outcomes in women undergoing in vitro fertilization (IVF). Follicular fluid and serum melatonin levels, oocyte quality, embryo development, and pregnancy rates were assessed.

DETAILED DESCRIPTION:
Background: Melatonin, a potent antioxidant, has been proposed to improve ovarian response and oocyte quality in assisted reproductive technologies (ART). This study evaluated the effects of melatonin supplementation on follicular fluid melatonin levels, hormonal profiles, and reproductive outcomes in women undergoing in vitro fertilization (IVF).

Methods: In this double-blind, randomized controlled trial, 80 infertile women were allocated to receive either 5 mg melatonin nightly (n=40) or placebo (n=40) during ovarian stimulation. Follicular fluid and serum melatonin levels, oocyte quality, embryo development, and pregnancy rates were assessed. Statistical analyses included Mann-Whitney U tests for continuous variables and chi-square/Fisher's tests for categorical data.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women aged 18-40 years
* No previous infertility treatment
* No previous hormonal treatment
* No previous radio-chemotherapy treatment

Exclusion Criteria:

* Fertile women
* Previous hormonal treatment
* Previous radio-chemotherapy treatment

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Follicular fluid melatonin concentration | Baseline (pre-intervention), periprocedurally and in the end of treatment at 7 weeks

SECONDARY OUTCOMES:
Reprodutive outcomes | From the enrollment to the end of treatment at 7 weeks
  (1) oocyte maturation rate (MII/oocytes retrieved), (2) blastocyst formation rate, (3) implantation rate (gestational sacs per embryo transferred), and (4) clinical pregnancy rate (ultrasound-confirmed at 7 weeks).

CONTACTS AND LOCATIONS:
Locations (1):
- Univertity of Sao Paulo, Clinics Hospital, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jamilian M, Foroozanfard F, Rahmani E, Talebi M, Bahmani F, Asemi Z. Effect of Two Different Doses of Vitamin D Supplementation on Metabolic Profiles of Insulin-Resistant Patients with Polycystic Ovary Syndrome. Nutrients. 2017 Nov 24;9(12):1280. doi: 10.3390/nu9121280. PMID 29186759
- [Result] Kloss JD, Perlis ML, Zamzow JA, Culnan EJ, Gracia CR. Sleep, sleep disturbance, and fertility in women. Sleep Med Rev. 2015 Aug;22:78-87. doi: 10.1016/j.smrv.2014.10.005. Epub 2014 Oct 18. PMID 25458772
- [Result] Fernando S, Rombauts L. Melatonin: shedding light on infertility?--A review of the recent literature. J Ovarian Res. 2014 Oct 21;7:98. doi: 10.1186/s13048-014-0098-y. PMID 25330986
- [Result] Schwertner A, Conceicao Dos Santos CC, Costa GD, Deitos A, de Souza A, de Souza IC, Torres IL, da Cunha Filho JS, Caumo W. Efficacy of melatonin in the treatment of endometriosis: a phase II, randomized, double-blind, placebo-controlled trial. Pain. 2013 Jun;154(6):874-81. doi: 10.1016/j.pain.2013.02.025. Epub 2013 Mar 5. PMID 23602498
- [Result] Ruder EH, Hartman TJ, Blumberg J, Goldman MB. Oxidative stress and antioxidants: exposure and impact on female fertility. Hum Reprod Update. 2008 Jul-Aug;14(4):345-57. doi: 10.1093/humupd/dmn011. Epub 2008 Jun 4. PMID 18535004
- [Result] Reiter RJ, Mayo JC, Tan DX, Sainz RM, Alatorre-Jimenez M, Qin L. Melatonin as an antioxidant: under promises but over delivers. J Pineal Res. 2016 Oct;61(3):253-78. doi: 10.1111/jpi.12360. Epub 2016 Sep 1. PMID 27500468
- [Result] Vander Borght M, Wyns C. Fertility and infertility: Definition and epidemiology. Clin Biochem. 2018 Dec;62:2-10. doi: 10.1016/j.clinbiochem.2018.03.012. Epub 2018 Mar 16. PMID 29555319